CLINICAL TRIAL: NCT04257916
Title: Effectiveness of Manual Therapy, Kinesiotape and Strength Training in Improving the Range of Ankle Movement, Stability, Strength and Pain in Soccer Players With Recurrent Ankle Sprains
Brief Title: Manual Therapy, Kinesiotape and Strength Training in Soccer Players With Recurrent Ankle Sprains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KTISO
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Ankle Sprains
Keywords: Kinesiotape; Myofascial; Ankle sprain; Pain; Stability
MeSH Terms: conditions — Ankle Injuries; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention by kinesiotape will be done with the player in supine position with the foot in dorsal flexion, anchoring the strip below the sole of the foot without tension, adding 50-70% tension until internal and external malleolus, and ending without tension. Another strip will be placed under the external malleolus, anchoring the bandage and following the talus (50-70% tension), leaving the scaphoid bulge free, surrounding the plant without tension and leaving the 5th metatarsal free. The bandage continues on the peroneal-astragalin ligament and the external malleolus (50-70% tension), until the tendon without tension. In the end we will surround the internal malleolus to the Achilles tendon without tension, ending with the same tension in the external malleolus and the neck of the talus.
  The myofascial technique and strength training will be the same in both groups.
  Interventions: Other: Experimental
- Control group (Active Comparator): The myofascial technique will be carried out by positioning the caudal hand of the physiotherapist in the astragalin and heel region, and the cranial hand in the middle foot. With a tibiotarsal traction, the foot will be everted, performing a shear in the astragalin zone, using a combined and slow technique.
  All players will warm up for 10 minutes on tape, at a speed of 7 km / h without inclination. The strength work was carried out with an isoinertial machine (Space Whell) with intervalic methodology: 20 "-10", with 4 series and doing three exercises: Squat, Lunges and Deadlift. One minute breaks will be made between sets.
  Interventions: Other: Manual therapy group

INTERVENTIONS:
Other: Experimental — Myofascial technique intervention of the subastragalar joint, kinesiotape and eccentric training with isoinercial machine. The intervention lasted 4 weeks. Each treatment session lasted 50 minutes, with 2 sessions a week. Between training sessions, the indicated break was 48 hours.
  Other Names: kinesio group
  Arms: Experimental group
Other: Manual therapy group — Myofascial technique of the subastragalar joint and eccentric training with isoinercial machine. The intervention lasted 4 weeks. Each treatment session lasted 50 minutes, with 2 sessions a week. Between training sessions, the indicated break was 48 hours.
  Arms: Control group

SUMMARY:
Introduction. The ankle sprain is one of the most prevalent injuries in soccer players. The muscle strength deficit is one of the variables that can most influence the development of a sprain. It has been indicated how the Kinesiotape and the myofascial direct induction technique can improve functionality.

Aim. To verify the effectiveness of the KinesioTape and the myofascial technique combined with strength training, in the reduction of pain, Rom increase, stability and strength in subjects who suffered ankle sprains.

Study design. Randomized, multicentric clinical study with follow-up. Methods. A random assignment of the subjects recruited in two study groups will be carried out: experimental and control group. The treatment will last 4 weeks, with 2 weekly sessions, of 50-60 minutes. The intervention includes the application of kinesiotape and myofascial treatment with strength training. The study variables will be pain (VAS), mobility (goniometer), stability (ProKin balance) and strength (MicroFet). A descriptive statistical analysis will be carried out calculating the main statistical characteristics. By means of the Kolmogorov-Smirnov test the distribution of the normality of the sample will be assessed. With the t-student test for related samples we will calculate the difference of means between the evaluations made in both groups. With an ANOVA of repeated measures we will calculate the intra and intersubject effect. The calculation of the effect size will be done with the Cohen formula.

Expected results. Improvement in stability, increase in range of motion, decrease in pain and increase in strength.

ELIGIBILITY:
Inclusion Criteria:

* Male soccer players
* 18 to 35 years old
* History of ankle sprain recurrences

Exclusion Criteria:

* Players who suffered a sprain in the previous month
* Footballers who were taking anti-inflammatory drugs
* Players undergoing another type of physiotherapy treatment at the time of the study
* Soccer players who do not sign the informed consent document.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline ankle range of motion after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done with a digital goniometer (Get my Rom model - Iphone 5 - Interactive Medical Productions). The movements of dorsal and plantar flexion, inversion and eversion will be measured. In measuring dorsal and plantar flexion, the goniometer will be placed on the 5th metatarsal. In measuring the inversion and eversion, the goniometer will be placed in the plantar part in line with the metatarsals. The unit of measure is the degree.

SECONDARY OUTCOMES:
Change from baseline isometric ankle strength after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A digital dynamometer (MicroFet®2 model - Hoggan Health Industries) will be used. To measure dorsal flexion, the instrument will be placed in the dorsal part of the foot in the region of the metatarsals, and for plantar flexion in the plantar part at the level of the metatarsals. In the eversion and abduction movements, the instrument will be placed in the lateral portion of the 5th metatarsal, while for inversion and adduction in the medial portion of the 1st metatarsal. Each movement will be repeated three times, one minute break.
Change from baseline stability after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done with the PWalk instrument. The software will allow measurement for 30 seconds with eyes open and closed. This measuring instrument will allow to evaluate: the movement with respect to the center of pressure in the frontal plane and sagittal plane (measured in mm). The evaluation will be done in charge.
Change from baseline ankle joint pain perception after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Pain assessment will be assessed through the visual analogue scale (VAS). Anteroposterior and mediolateral movements will be performed. This scale is used using a scale of 0 to 10 points, where 0 indicates no pain and unstable, 10 indicates the maximum pain perceived.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- European University of Madrid, Madrid, Spain